CLINICAL TRIAL: NCT06155929
Title: Traveler's Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Sebastian Hansen, Medical student, Herlev Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: F-23025419
Record Dates: First submitted 2023-04-27; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Constipation; Travel-Related Illness
MeSH Terms: conditions — Constipation; Travel-Related Illness

STUDY DESIGN:
Intervention Model Description: The investigators are investigating wether a flight abroad is causing a decrease in stools.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Flight (Other): The intervention is the flight to turkey and home to Denmark again.
  Interventions: Behavioral: Flight

INTERVENTIONS:
Behavioral: Flight — The participants are flying to turkey and back home. The flights are the intervention.

SUMMARY:
The occurence of traveler's constipation is sparsely covered in the medical litterature. This study aims to determine the gastrointestinal-related discomforts related to traveling on a trip to Turkey.

DETAILED DESCRIPTION:
Traveler's constipation, which is characterized by the more hard and less frequent stools, is sparsely covered in the medical litterature. Only a few studies have examined this problem and the actual occurrence and extent of this problem is not known. Hypotheses about why travel constipation occurs are, among other things, about changed circadian rhythm due to jet lag, changed schedules and tight sanitary conditions. Other factors such as dehydration, change in cabin pressure and the content of the in-flight food in connection with flights have not been investigated.

The research project aims to clarify changes in the test subjects' bowel habits as well as other gastrointestinal-related discomforts in connection with a flight abroad with only an hour's time difference and without the consumption of flight food.

ELIGIBILITY:
Inclusion Criteria:

* Can understand danish and is able to answer the questionnaires
* Given written consent

Exclusion Criteria:

* History of intestinal resection
* Medically treated intestinal disease
* IBS at baseline

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
Stool frequency | 14 days
  The investigators are sending questionnaires to the participants of the study to decide wether the stool frequency decreases after flight to turkey. No scale used, simply time and number.

SECONDARY OUTCOMES:
Bristol Stool Chart. | 14 days
  The investigators are evaluating if the stool becomes less liquid indicating a prolonged transition time. On er Likert scale from 1-7, 7 being most wet.
VAS-IBS: Visual Analog Scale for Irritable Bowel Syndrome | 14 days
  Scale from 0-100 describing gastrointestinal bloating, pain and discomfort. 0 being good and 100 being bad

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev Hospital, Herlev, Danmark, Denmark

IPD SHARING:
Plan to Share IPD: No